CLINICAL TRIAL: NCT00785499
Title: The Effect of Milk, Whey and Casein on Weight Loss and Risk Markers of Metabolic Syndrome in Overweight Children
Brief Title: Milk Components and Metabolic Syndrome
Acronym: MoMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, AAstrup, Prof, University of Copenhagen
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: MoMS D204
Record Dates: First submitted 2008-11-04; First posted 2008-11-05 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Obesity; Metabolic Syndrome
Keywords: obesity; metabolic syndrome; milk components; casein; whey; children; adolescent
MeSH Terms: conditions — Obesity; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- skim milk (Experimental): skim milk
  Interventions: Behavioral: Milk Components and Metabolic syndrome
- whey (Experimental): Whey milk drink
  Interventions: Behavioral: Milk Components and Metabolic syndrome
- casein (Experimental): casein milk drink
  Interventions: Behavioral: Milk Components and Metabolic syndrome
- water (Active Comparator): Danish mineral water
  Interventions: Behavioral: Milk Components and Metabolic syndrome

INTERVENTIONS:
Behavioral: Milk Components and Metabolic syndrome — 1 liter per day of the test drinks for 3 mo

SUMMARY:
Milk contains a vast number of bioactive components that have been suggested to have a positive impact on human health, of special interest is the effects related to metabolic syndrome and obesity but the effect of the individual milk components is not clear. This study examine whether it is beneficial for overweight and obese children to increase the intake of skim milk, or whey or casein in relation to bodyweight and markers of MS.

The participants will be randomized to receive skim milk, whey milk drink, casein milk drink or mineral water for 3 mo. They will be examined at baseline, end of intervention and followed up 3 month later.

ELIGIBILITY:
Inclusion Criteria:

* 12 years to 15 years old
* iso BMI larger than 25
* habitual milk intake less than 250 ml/day
* non-smoker
* healthy at the time of inclusion

Exclusion Criteria:

* chronic illnesses
* intake of antibiotic 1 mo before start of intervention

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 193 (Actual)
Dates: Start 2008-11; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
body composition and markers for metabolic syndrome (e.g.fasting insulin, glucose, lipid profile, CRP, PAI-1, tPA) | at baseline, after intervention and body composition 3 mo after end of intervention

SECONDARY OUTCOMES:
diet | baseline and end of intervention
pulse wave velocity, | baseline and end of intervention
blood pressure, metabolomics, IFG-I, IGFBP-3, appetite regulatory hormones,immune parameters, bone turn over parameters, composition of microbiota, vitamin D, physical activity | baseline and end of intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Human Nutrition, Frederiksberg, Denmark

REFERENCES:
- [Derived] Andersen LB, Arnberg K, Trolle E, Michaelsen KF, Bro R, Pipper CB, Molgaard C. The effects of water and dairy drinks on dietary patterns in overweight adolescents. Int J Food Sci Nutr. 2016;67(3):314-24. doi: 10.3109/09637486.2016.1150435. Epub 2016 Feb 22. PMID 26903408
- [Derived] Arnberg K, Molgaard C, Michaelsen KF, Jensen SM, Trolle E, Larnkjaer A. Skim milk, whey, and casein increase body weight and whey and casein increase the plasma C-peptide concentration in overweight adolescents. J Nutr. 2012 Dec;142(12):2083-90. doi: 10.3945/jn.112.161208. Epub 2012 Oct 17. PMID 23077192
- [Derived] Arnberg K, Larnkjaer A, Michaelsen KF, Molgaard C. Central adiposity and protein intake are associated with arterial stiffness in overweight children. J Nutr. 2012 May;142(5):878-85. doi: 10.3945/jn.111.150672. Epub 2012 Mar 21. PMID 22437560